CLINICAL TRIAL: NCT02000128
Title: A Prospective, Randomized Controlled Study of Bioimpedance Analysis(BIA) Guided Fluid Management in Peritoneal Dialysis Patients.
Brief Title: Fluid Management Guided by Bioimpedance Analysis in Peritoneal Dialysis(PD) Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Director, Institute of Nephrology, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PD-BIA
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: End Stage Renal Disease
Keywords: Peritoneal Dialysis; fluid overload; bioimpedance analysis; Randomized Controlled Trial
MeSH Terms: conditions — Kidney Failure, Chronic; Edema | interventions — Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bioimpedance monitoring group (Experimental): patients whose fluid status will be monitored and guided by bioimpedance analysis
  Interventions: Device: bioimpedance monitoring
- clinical monitoring group (Other): patients whose fluid status will be monitored and guided by clinical experience
  Interventions: Other: clinical monitoring

INTERVENTIONS:
Device: bioimpedance monitoring — To assess the body composition using Multi-frequency bioelectrical impedance analysis
  Other Names: Multi-frequency bioelectrical impedance analysis; Body Composition Analyzer
  Arms: bioimpedance monitoring group
Other: clinical monitoring — clinical symptom and examination,such as edema, body weight, blood pressure, cardial function
  Other Names: routine method of assessing water status
  Arms: clinical monitoring group

SUMMARY:
1. Purpose: to investigate the effect of bioimpedance analysis(BIA) guided fluid management versus experiential way on clinical outcome in peritoneal dialysis patients.
2. Design: prospective,randomized,controlled,single center study
3. Study hypothesis: Patients on peritoneal dialysis are frequently hypervolemic, which is associated with increasing hazard of death and cardiovascular events. Bioimpedance analysis is a safe, and easy way, which appears to be more useful and sensitive than other techniques for assessing volume status in dialysis patients. Therefore we hypothesize that more concise and strict fluid management guided by BIA may help to improve patients' survival, decrease cardiovascular events and hospitalization rate.
4. Objects: incident and prevalent patients with overhydration status.

   1. anticipated cases:240
   2. arms: all the patients are randomized into two arms.(BIA group/clinical group)
   3. observational time:12 months
5. Primary Outcome: all cause mortality. Secondary Outcomes: technique survival, cardiovascular events, peritonitis, residual renal function.

ELIGIBILITY:
Inclusion Criteria:

* patients who are undergoing peritoneal dialysis and clinically stable for at least 3 months;
* 18 Years and older;
* ratio extracellular water (ECW)/total body water(TBW)≧0.4;
* signed the informed consent

Exclusion Criteria:

* patients who have mental graft;
* amputation;
* patients who is unable to accomplish the BIA measurement in standing position for 3 minutes;
* patients whose heart function are class IV estimated by New York Heart Association (NYHA) standard;
* Patients who have acute complications within 30 days prior to study enrollment;
* patients whose life expectancy is within 6 months;
* patients who are pregnant;
* patients who are unable to give consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
death | 12 months
  all cause mortality;cardiovascular related mortality

SECONDARY OUTCOMES:
technique failure | 12 months
  permanent hemodialysis transfer
cardiovascular events | 12 months
  heart failure, myocardial infarction,angina, Percutaneous coronary stenting, coronary artery bypass grafting,
clinical adverse events | 12 months
  hospitalization events due to overload; Non-PD related infection; PD related peritonitis; peripheral angiopathy
residual renal function | 12 months
  change of baseline residual renal function, measured as residual glomerular filtration rate(rGFR) and urine volume

CONTACTS AND LOCATIONS:
Overall Officials: Xuqing Yu, MD,PHD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China